CLINICAL TRIAL: NCT01718340
Title: Phase 4 Study of Effectiveness of Metformin in Patients With Unexplained Recurrent Miscarriages
Brief Title: Effectiveness of Metformin in Recurrent Miscarriage in a Woman With Hyperinsulinaemia
Acronym: MetRPL
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, alaa eldeen mahmoud ismail, M D, Woman's Health University Hospital, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MetRPL
Record Dates: First submitted 2012-08-18; First posted 2012-10-31 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Abortion, Habitual
Keywords: PCOS; Hyper insulinaemia; metformin; recurrent abortion
MeSH Terms: conditions — Abortion, Habitual | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): The patients with PCO and hyper insulinemia will be subdivided into two groups, one group will continue metformin 500 mg three times per day from the start of induction of ovulation till the end of pregnancy, the other group will stop the drug once pregnancy test become positive
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — metformin tablet 500mg three time per day
  Other Names: glucophage; cidophage; amophage

SUMMARY:
The prevalence of insulin resistance is increased in women with recurrent miscarriage compared with matched fertile controls,Insulin resistance (IR) in this syndrome is not only implicated toward early pregnancy loss (EPL) but also pathognomic for various obstetrical complications during pregnancy.An elevated free androgen index appears to be a prognostic factor for a subsequent miscarriage in women with recurrent miscarriage.

There is insufficient evidence to evaluate the effect of metformin supplementation in pregnancy to prevent a miscarriage in women with recurrent miscarriage.

DETAILED DESCRIPTION:
The patients with PCO and hyper insulinemia will be subdivided into two groups, one group will continue metformin 500 mg three times per day from the start of induction of ovulation till the end of pregnancy, the other group will stop the drug once pregnancy test become positive. Pregnancy follow up including the early and second trimester pregnancy loss, Secondary outcomes like gestational diabetes, pregnancy-induced hypertension and intrauterine growth restriction were also analyzed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* women who are diagnosed to have PCOS and/or haven hyper insulinaemia and have a previous history of recurrent miscarriages.

Exclusion Criteria:

* Any patients with PCOS or hyper insulinaemia previously treated by any forms of insulin sensitizers.

Age above forty years old .

* Antiphospholipid syndrome (lupus anticoagulant and/or anticardiolipin antibodies [IgG or IgM]); other recognised thrombophilic conditions (testing according to usual clinic practice).
* Intrauterine abnormalities (as assessed by ultrasound, hysterosonography, hysterosalpingogram, or hysteroscopy).
* Fibroids distorting uterine cavity .
* Abnormal parental karyotype .
* Other identifiable causes of recurrent miscarriages (tests initiated only if clinically indicated) e.g., diabetes, thyroid disease and systemic lupus erythematosus (SLE).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to evaluate the clinical pregnancy rate and the effectiveness of Metformin in the reduction of EPL in women with PCOS | 2 ys
  The patients with PCO and hyper insulinemia will be subdivided into two groups, one group will continue metformin 500 mg three times per day from the start of induction of ovulation till the end of pregnancy,

SECONDARY OUTCOMES:
Secondary outcomes like gestational diabetes, pregnancy-induced hypertension and intrauterine growth restriction were also analyzed at the end of the study and any fetal malformation | 2 ys
  The patients with PCO and hyper insulinemia will be subdivided into two groups, one group will continue metformin 500 mg three times per day from the start of induction of ovulation till the end of pregnancy, the other group will stop the drug once pregnancy test become positive. Pregnancy follow up including the early and second trimester pregnancy loss, Secondary outcomes like gestational diabetes, pregnancy-induced hypertension and intrauterine growth restriction were also analyzed at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Ismail, M D, Principal Investigator — Faculty of medicine,Assiut university,Egypt
Locations (1):
- Women's Health Hospital, Asyut, Egypt